CLINICAL TRIAL: NCT00324584
Title: Surveillance Des données De l'Autosurveillance glycémique Via Internet Et Le réseau téléphonique GSM Chez Le diabétique De Type 1 Sous Traitement Insulinique Par Pompe Externe : Etude Prospective randomisée PumpNet.
Brief Title: Web-Based Follow-Up Using Cellular Phone in Type 1 Diabetic Patients Under Insulin Pump Therapy : The PumpNet Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Grenoble (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: DCIC 03 01
Record Dates: First submitted 2006-05-10; First posted 2006-05-11 (Estimated); Last update posted 2006-07-07 (Estimated); Status verified 2006-07

CONDITIONS: Type 1 Diabetes Mellitus
Keywords: type 1 diabetes mellitus; telecare; telemedicine; insulin pump therapy
MeSH Terms: conditions — Diabetes Mellitus, Type 1

INTERVENTIONS:
Device: Telemonitoring of glucose values using GlucoNet device

SUMMARY:
The purpose of this study is to determine if telecare using modern telecommunication devices can improve the metabolic control and the quality of life of type 1 diabetic patients.

DETAILED DESCRIPTION:
We aim at comparing conventional follow-up of type 1 diabetic patients treated with continuous subcutaneous insulin infusion (CSII) (face-to-face visits) with an intensive coaching using the Web and the cellular phone network for data transmission and Short Message Service (SMS). This telecommunication device is called GlucoNet. The specific objectives are to measure the efficiency of GlucoNet in improving metabolic control, reducing health care costs and improving the quality of life of patients.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 diabetes mellitus
* Age ≥ 18
* HbA1c between 7.5 and 10%
* Treated with continuous subcutaneous insulin infusion for a minimum of 3 months

Exclusion Criteria:

* Unstabilized diabetic microangiopathy
* Ongoing pregnancy or planned pregnancy
* Unwilling to perform a minimum of 4 capillary blood tests per day
* Unable to use the GlucoNet device

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40
Dates: Start 2003-04; Study Completion 2004-09

PRIMARY OUTCOMES:
Glycated hemoglobin HbA1c
monthly mean capillary blood glucose value
blood glucose variability index (MAGE Index and LBGI index)
quality of life score (DQOL score)
frequency of hypoglycemic episodes (<70 mg/dl)

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Y Benhamou, MD, PhD, Principal Investigator — Universty Hospital, Grenoble, France; Helene Hanaire, MD, PhD, Study Director — University Hospital, Toulouse, France; Serge Halimi, MD, Study Director — University Hospital, Grenoble, France; Jean L Bosson, MD, PhD, Study Director — CIC-INSERM
Locations (2):
- France (2):
  - University Hospital, Department of Endocrinology, Grenoble
  - University Hospital, Department of Endocrinology, Toulouse